CLINICAL TRIAL: NCT03226951
Title: Sub Threshold Laser for Non Central Diabetic Clinical Significant Macular Edema
Brief Title: SDM Laser for Non Central Diabetic CSME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marashi Eye Clinic (Other)
Responsible Party: Principal Investigator, Ameen Marashi, Principle investigator, Marashi Eye Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol DME 2
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Non Central Diabetic Macular Edema
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subtherhold 532 nm laser (Experimental): Applying 532nm subtherhold laser with 5% duty cycle using high density low intensity protocol at the area of non central clinical significant macular edema
  Interventions: Device: Subthreshold 532nm laser

INTERVENTIONS:
Device: Subthreshold 532nm laser — Subthershold 532nm laser

SUMMARY:
Is to determine if SDM laser can reduce macular thickness in non central CSME and stop the progression of non central CSME to central CSME in compare to glycemic control

DETAILED DESCRIPTION:
interventional randomised masked study will recruit patients have diabetes mellitus with non central CSME with good vision into two groups : 1st SDM laser with glycemic control 2nd SHAM laser with Glycemic control where BCVA will be recorded every month starting from baseline to 24 weeks where OCT will be recorded every 8 weeks from baseline to 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients with central diabetic macular edema Best corrected visual acuity is 20/30 or more
* Non central Macular thickness more than 250 microns
* Patients who are able to come for all follow-up

Exclusion Criteria:

* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 3 years.
* Macular edema is present that is considered to be related to ocular surgery such as cataract extraction
* Substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by 3 lines or more
* History of major ocular surgery (including vitrectomy, scleral buckle, any intraocular surgery, etc.) within prior 4 months or anticipated within the next 6 months following randomization.
* Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Number of eyes with reduced macular thickness | 24 weeks
  Measurements of retinal thickness in the area of edema

SECONDARY OUTCOMES:
Number of eyes with reduced vision | 24 weeks
  Best corrected visual acuity at the end of the study
Number of eyes developing central macular edema | 24 weeks
Number of patients achieved good glycemic control | 24 weeks
  By measuring HbA1C every 12 weeks from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Marashi Eye Clinic, Aleppo, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marashi A. Non-central diabetic clinical significant macular edema treatment with 532nm sub threshold laser. Adv Ophthalmol Vis Syst. 2018;8(3):151-154. DOI: 10.15406/aovs.2018.08.0029
- See also: Non-central diabetic clinical significant macular edema treatment with 532nm sub threshold laser — http://medcraveonline.com/AOVS/AOVS-08-00291.pdf